CLINICAL TRIAL: NCT01581723
Title: Using Biploar Technology for Transurethral Resection of Bladder Tumor - a Randomized Controlled Trial
Brief Title: Clinical Trial Using Bipolar Technology for Transurethral Resection of Bladder Tumor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Eddie SY Chan, MD, Dr., Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUHK_TURB_2012
Record Dates: First submitted 2012-03-21; First posted 2012-04-20 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Urinary Bladder Tumor
Keywords: urinary bladder tumor; monopolar TURBT; bipolar TURBT
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monopolar TUR (Active Comparator): Monopolar diathermy is used to perform tranurethral resection of bladder tumor
  Interventions: Device: Monopolar diathermy
- Biploar TUR (Experimental): Bipolar diathermy is used to perform transurethral resection of bladder tumor
  Interventions: Device: Bipolar diathermy

INTERVENTIONS:
Device: Monopolar diathermy — monopolar diathermy
  Other Names: Olympus Monopolar HF-resection Electrode; Model: A22205A
  Arms: Monopolar TUR
Device: Bipolar diathermy — bipolar diathermy
  Other Names: Olympus TURis Bipolar HF-resection electrode; Model: WA22306D
  Arms: Biploar TUR

SUMMARY:
Bladder cancer is a common urological malignant disease. Patients with bladder cancer will first be managed with transurethral resection (TUR) of bladder tumor. For many years, monopolar transurethral resection of bladder tumor (TURP) has been the gold standard for treatment. However, complications including bleeding, bladder perforation and inadequate sampling of deep tumor biopsy remain the major concerns. Recently published papers suggested that the newer bipolar TUR technology has similar surgical outcomes but less complications comparing with monopolar TUR. In this study, investigators will investigate the benefit of new technology as compared with conventional monopolar resection on tumor clearance, complication and recurrence rates.

DETAILED DESCRIPTION:
Transurethral resection (TUR) of bladder tumor is one of commonest procedures in urology practice. It is the surgery of choice for staging and treating non-muscle invasive bladder cancer. Short lengths of hospital stay, simple and safe are the main advantages of the surgery. Conventional TUR is performed with monopolar diathermy, which commonly elicits obturator reflexes in lateral-located tumor. However, it is not without complication. Bleeding and bladder perforation with or without obturator reflex are the most significant complications after TUR of bladder tumor. The charring effect of monopolar is also a concern as the diagnosis of muscle invasion by tumor is determined by the integrity of tumor base biopsy. Mariappan et al. reported that as high as 33% of the specimen had no detrusor muscle present for assessment. The absent of muscle not only affect the staging procedure but also associated with higher cancer recurrence rate.

Bipolar resection has been widely used in transurethral resection of prostate (TURP). As compared with the traditional monopolar technology, the electric current passes through the instrument sheath. The advantage of bipolar technology includes less obturator reflex, good hemostasis and early recovery. Study has showed that the cautery artifact is more severe on monopolar resection as compared with bipolar in prostate tissues. Due to the clean and precise cutting, there will be less charring on the specimen and thermal injury to peripheral tissues. Applying to bladder tumor resection, this will improve the staging accuracy with better determination of the depth of invasion. Furthermore, with the use of saline instead of glycine as irrigation fluid, risk of TUR syndrome is minimized. There is no randomized trial on the benefit of using bipolar instrument on TUR bladder cancer. In this study, investigator will investigate the role of bipolar technology in TUR bladder cancer as compared with traditional monopolar resection.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients (age ≥ 18)
* Patients who have diagnosed with bladder cancer (either primary or recurrent) by cystoscopy

Exclusion Criteria:

* Patients who are scheduled for second TUR within 6 weeks after the previous TUR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Muscle sampling rate | An expected average of 7 days post operation
  To assess the charring effect to the integrity of the tumor base biopsy
Incidence of TUR syndrome | Intra-operation and up to 7 days post operation

SECONDARY OUTCOMES:
Recurrence rate of bladder cancer | 3 months and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eddie SY Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin
  - North District Hospital, Sheung Shui